CLINICAL TRIAL: NCT04365114
Title: Patient Outcomes from Second Film-readers and Test Threshold Relaxation in Breast Screening: an Observational Retrospective Cohort Study
Brief Title: Patient Outcomes from Second Film-readers and Test Threshold Relaxation in Breast Screening
Acronym: POSTBOx
Status: Completed | Type: Observational
Sponsor: University of Warwick (Other)
Collaborators: Public Health England (Other Government)
Responsible Party: Principal Investigator, Sian Taylor-Phillips, Associate Professor of Screening and Test Evaluation, University of Warwick
Other Study IDs: 50619
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Ductal Carcinoma in Situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Speech Reception Threshold Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Single reading: Only one clinician examined the woman's mammograms for signs of cancer and recommended whether to recall her for further tests or not.
  Interventions: Diagnostic Test: Breast Screening Mammography with single reader; Diagnostic Test: Test threshold
- Double reading: Two clinicians examined the woman's mammograms for signs of cancer and recommended whether to recall her for further tests or not.
  Interventions: Diagnostic Test: Breast screening mammography with two readers; Diagnostic Test: Test threshold

INTERVENTIONS:
Diagnostic Test: Breast Screening Mammography with single reader — One clinician examined each woman's mammograms for signs of cancer
  Groups: Single reading
Diagnostic Test: Breast screening mammography with two readers — Two clinicians seperately examined each woman's mammograms for signs of cancer
  Groups: Double reading
Diagnostic Test: Test threshold — Threshold used by readers examining the breast screening mammograms, defined using their previous proportion of cases recalled

SUMMARY:
Analysis of women's medical records to understand the impact of previous changes to breast cancer screening (increase from one to two clinicians examining each woman's mammograms, and what proportion of women they recall for further tests)

DETAILED DESCRIPTION:
Retrospective observational study examining the records and outcomes of women who attended breast cancer screening between 1988 and 2016. Linkage of records from the breast screening service, the cancer registry, and mortality. Analysis of whether changing the threshold for whether to recall women for further tests or the number of clinicians examining the mammograms for signs of cancer affects outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women who attended the English National Health Service (NHS) breast cancer screening service at least once between 1988 and 2016, aged between 47 and 73
* All eligible episodes of screening for each woman (we expect women to be screened around 7 times each)

Exclusion Criteria:

* Women who did not attend routine English NHS Breast screening service within the specified date and age range, even if they attended symptomatic breast cancer services, high risk (family history) breast screening services, or if they were referred for mammograms by their general practitioner

Ages: 47 Years to 73 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who attended the English NHS Breast screening programme between 1988 and 2016 aged between 47 and 73.
Sampling Method: Probability Sample
Enrollment: 13094122 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Number of women overdiagnosed (the cancer would not have become symptomatic within the woman's lifetime) using compensatory drop method | 13 years, and up to 30 years
  Overdiagnosis of breast cancer (measured as difference in total cancer incidence, screen and symptomatic). Will also report mechanism of action (number of screen detected cancers, number of symptomatically detected cancers at 3,13, and 30 years follow-up)
Cancers detected at screening | 1 day screening episode
  Biopsy proven cancers detected at screening
False positive recalls | 1 day screening episode
  Recall of women for further tests after screening which did not result in detection of cancer
Breast cancer mortality | 13 years, and up to 30 years
  Mortality due to breast cancer (dependent on securing follow-on funding)
All cause mortality | 13 years, and up to 30 years
  Mortality due to any cause (dependent on securing follow on funding)
Characteristics of cancer detected | 1 day screening episode, 3year, 13 year and up to 30 year follow up
  Size, grade and stage (reported overall, screen detected, and symptomatic detected).

SECONDARY OUTCOMES:
Breast cancer morbidity | Up to 30 years
  Treatment received as a proxy for treatment associated morbidity (reported overall, screen detected and symptomatically detected, if follow on funding obtained)
Breast cancer free survival | Up to 30 years follow-up
  Survival without a diagnosis of breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Sian Taylor-Phillips, PhD, Principal Investigator — University of Warwick
Locations (1):
- Univesity of Warwick, Coventry, Warwickshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We do not have Office of Data Release permissions to share these data with other researchers

REFERENCES:
- See also: Study website — https://warwick.ac.uk/fac/sci/med/research/hscience/pet/projects/postbox